CLINICAL TRIAL: NCT00743132
Title: Novel Prediction Score for Postoperative Acute Renal Failure (ARF) Following Liver Resection
Acronym: StV 11-2008
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: med. pract. Ksenija Slankamenac, Swiss HPB (Hepato-Pancreato-Biliary) Center, Department of Surgery
Other Study IDs: StV 11-2008; StV 11-2008
Record Dates: First submitted 2008-08-27; First posted 2008-08-28 (Estimated); Last update posted 2010-01-25 (Estimated); Status verified 2010-01

CONDITIONS: Acute Renal Failure
Keywords: evaluation; incidence; liver surgery; resection; impact; postoperative; mortality
MeSH Terms: conditions — Acute Kidney Injury; Tooth, Impacted

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Postoperative no renal dysfunction
- 2: Postoperative renal dysfunction

SUMMARY:
ARF is a frequent event after hepatic resection and therefore clinically highly relevant.

There is limited evidence on the incidence of postoperative ARF and its clinical relevance in patients undergoing liver resection.

This study will evaluate the incidence of acute renal failure (ARF) after liver resection and its impact on postoperative mortality.

DETAILED DESCRIPTION:
ARF is a frequent event after hepatic resection and therefore clinically highly relevant.

There is limited evidence on the incidence of postoperative ARF and its clinical relevance in patients undergoing liver resection.

This study will evaluate the incidence of acute renal failure (ARF) after liver resection and its impact on postoperative mortality.

ELIGIBILITY:
Inclusion Criteria:

* Patient age >/= 18 years
* Benign and malign liver diseases

Exclusion Criteria:

* Trauma cases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with benign and malign liver diseases of the Swiss HPB (Hepato-Pancreato-Biliary) Center undergoing liver resection from 2002 - 2007
Sampling Method: Non-Probability Sample
Enrollment: 569 (Actual)
Dates: Start 2008-04; Primary Completion 2008-10 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Predictor score
Incidence of ARF Length of hospital stay

CONTACTS AND LOCATIONS:
Locations (1):
- Swiss HPB (Hepato-Pancreato-Biliary) Center of the University Hospital Zurich, Zurich, Canton of Zurich, Switzerland

REFERENCES:
- [Derived] Slankamenac K, Breitenstein S, Held U, Beck-Schimmer B, Puhan MA, Clavien PA. Development and validation of a prediction score for postoperative acute renal failure following liver resection. Ann Surg. 2009 Nov;250(5):720-8. doi: 10.1097/SLA.0b013e3181bdd840. PMID 19809295